CLINICAL TRIAL: NCT02734862
Title: A Phase 2, Multicenter, Randomized, Double-blind Study of the Safety, Tolerability, and Efficacy of Intravenous CD101 vs Intravenous Caspofungin Followed by Oral Fluconazole Step-down in the Treatment of Subjects With Candidemia and/or Invasive Candidiasis
Brief Title: CD101 Compared to Caspofungin Followed by Oral Step Down in Subjects With Candidemia and/or Invasive Candidiasis-Bridging Extension
Acronym: STRIVE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cidara Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CD101.IV.2.03; 2015-005599-51 (EudraCT Number)
Record Dates: First submitted 2016-03-16; First posted 2016-04-12 (Estimated); Results first posted 2020-12-08 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: Candidemia; Mycoses; Fungal Infection; Fungemia; Invasive Candidiasis
Keywords: mycoses
MeSH Terms: conditions — Candidemia; Mycoses; Fungemia; Candidiasis, Invasive | interventions — Injections; Caspofungin; Fluconazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): Subjects in the CD101 IV treatment group 1 (Part A Only - up to 30 mITT subjects) will receive CD101 IV 400 mg on Day 1 and Day 8, with an optional dose of 400 mg on Day 15 (for all subjects) and an optional dose of 400 mg on Day 22 (only for subjects with IC), if needed.
  Daily intravenous placebo infusion when not administered CD101. Daily oral placebo as step down.
  Interventions: Drug: CD101; Drug: intravenous placebo; Drug: oral placebo
- Group 3 (Active Comparator): Subjects in the caspofungin group will receive IV caspofungin (a single 70 mg loading dose on Day 1 followed by 50 mg once daily) for ≥3 days up to a maximum of 21 days for subjects with candidemia only and up to a maximum of 28 days for subjects with IC (with or without candidemia).
  After ≥3 days of IV therapy, subjects in the caspofungin group can be switched to oral step-down therapy of fluconazole (a loading dose of 800 mg [4 capsules] on the first day followed by 400 mg [2 capsules]/day thereafter). After switch to oral step down before Day 8, subjects in the caspofungin group will receive IV placebo on Day 8 to preserve the study blind.
  Interventions: Drug: Caspofungin; Drug: Fluconazole; Drug: intravenous placebo
- Group 2 (Experimental): Subjects in the CD101 IV treatment group 2 (Part B Only - up to 30 mITT subjects) will receive CD101 IV 400 mg on Day 1 and Day 8, with an optional dose of 200 mg on Day 15 (for all subjects) and an optional dose of 200 mg on Day 22 (only for subjects with IC), if needed.
  Daily intravenous placebo infusion when not administered CD101. Daily oral placebo as step down.
  Interventions: Drug: CD101; Drug: intravenous placebo; Drug: oral placebo

INTERVENTIONS:
Drug: CD101 — Intravenous antifungal therapy
  Other Names: CD101 for Injection
  Arms: Group 1; Group 2
Drug: Caspofungin — Intravenous antifungal therapy
  Other Names: Cancidas
  Arms: Group 3
Drug: Fluconazole — oral antifungal therapy
  Other Names: generic fluconazole
  Arms: Group 3
Drug: intravenous placebo — normal saline
  Other Names: placebo infusion
Drug: oral placebo — microcrystalline cellulose
  Other Names: encapsulated cellulose
  Arms: Group 1; Group 2

SUMMARY:
The purpose of this study is to determine if intravenous CD101 is safe and effective in the treatment of candidemia and/or invasive candidiasis when compared to caspofungin (followed by oral fluconazole).

DETAILED DESCRIPTION:
This Bridging Extension is to determine if intravenous CD101 is safe [Day 45- 52 for subjects with candidemia only, or Day 52- 59 for subjects with invasive candidiasis with or without candidemia] and effective [Day 14 (± 1 day)] in the treatment of candidemia and/or invasive candidiasis when compared to caspofungin (followed by oral fluconazole).

ELIGIBILITY:
Inclusion Criteria:

* mycological diagnosis of candidemia and/or invasive candidiasis from a sample taken less than or equal to 96 hours before randomization (defined as: at least 1 blood culture positive for Candida or positive test for Candida from a sponsor approved rapid diagnostic test or positive gram stain for yeast or positive culture for Candida spp. from a specimen obtained from a normally sterile site)
* willing to initiate or continue medical treatment to cure infections, including receipt of antibiotics and surgical procedures, if required. Patients receiving only medications and measures for comfort and not cure should not be enrolled.
* female subjects of child bearing potential <2 years post menopausal must agree to one barrier method and one highly effective method of birth control or sexual abstinence.
* male subjects must be vasectomized, abstain from sexual intercourse, or agree to use barrier contraception (condom with spermicide), and also agree not to donate sperm from first dose of CD101 (Day 1) until 90 days following last administration of study drug.
* willing and able to provide written informed consent. If the subject is unable to consent for himself/herself, a legally acceptable representative must provide informed consent on their behalf.
* presence of one or more systemic signs attributable to candidemia and/or invasive candidiasis

Exclusion Criteria:

* Any of the following forms of IC:

  1. Septic arthritis in a prosthetic joint (septic arthritis in a native joint is allowed)
  2. Osteomyelitis
  3. Endocarditis or myocarditis
  4. Meningitis, endophthalmitis, or any central nervous system infection
* neutropenia
* alanine aminotransferase or aspartate aminotransferase levels >10 fold the upper limit of normal
* severe hepatic impairment in subjects with a history of chronic cirrhosis
* greater than 48 hours systemic antifungal treatment at approved doses to treat candidemia
* pregnant females
* lactating females who are nursing
* known hypersensitivity to CD101, caspofungin, any echinocandin, or to any of their excipients
* previous participation in this or any previous CD101 study
* recent use of an investigational medicinal product within 28 days of first dose of study drug or presence of an investigational device at the time of screening
* Principal Investigator considers the subject should not participate
* presence of indwelling vascular catheter or device that cannot be removed and is likely to be the source of candidemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2016-07-26 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Taylor Sandison, MD MPH, Study Director — Cidara Therapeutics
Locations (63):
- United States (16):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California - Davis, Davis, California
  - University of Miami Miller School of Medicine, Miami, Florida
  - Augusta University, Augusta, Georgia
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Harper University Hospital, Detroit, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Washington University School of Medicine, St Louis, Missouri
  - Mercury Street Medical, Butte, Montana
  - Albany Medical Center, Albany, New York
  - Mercy Health - St. Vincent Medical Center - ID Clinical Research, Toledo, Ohio
  - Reading Hospital and Medical Center, West Reading, Pennsylvania
  - University of Texas Health Science Center at Houston, Houston, Texas
  - Virginia Tech, Carillion School of Medicine, Roanoke, Virginia
- Belgium (8):
  - Jules Bordet Institute, Brussels
  - CHU Brugman, Brussels
  - Erasme Hospital, Brussels
  - UCL Saint-LUC, Brussels
  - UZ Gent Algemene Inwendige Zietken, Ghent
  - University Hospital Brussels, Jette
  - University Hospital Leuven, Leuven
  - CHU Sart-Tillman, Liège
- Bulgaria (2):
  - University Multiprofile Hospital for Active Treatment "Sveti Ivan Rilski", Sofia, Clinic of Clinical Hematology, Sofia
  - University Multiprofile Hospital for Active Treatment and Emergency Medicine "N.I. Pirogov", Sofia, Burns and Plastic Surgery Clinic, Department of Anesthesiology and Intensive Care, Sofia
- Canada (4):
  - Juravinski Hospital and Cancer Centre/Hamilton Health Sciences, Hamilton, Ontario
  - Toronto General Hospital-University Health Network, Toronto, Ontario
  - CIUSSS de L'Est-de-l'Île-De-Montréal, Installation Hôpital, Montreal, Quebec
  - McGill University Health Centre-Research Institute, Montreal, Quebec
- Greece (6):
  - University General Hospital "Attikon", 2nd Department of Critical Care, Athens, Chaidari
  - General Hospital of Athens "Evangelismos", 5th Department of Internal Medicine and Infectious Diseases Unit, Athens
  - Laiko General Hospital of Athens, Athens
  - Henry Dunant Hospital Center, Athens
  - General Hospital of Athens "Evangelismos", Department of Critical Care, Athens
  - University Hospital of Larissa, Department of Critical Care Unit, Thessaloniki
- Hungary (2):
  - Medical Centre, Hungarian Defence Forces, Central Intensive Care Unit and Anesthesiology Department, Budapest
  - Fejer County St. Gyorgy University Teaching Hospital, Central Department of Anesthesiology and Intensive Care Unit, Szeged
- Italy (6):
  - Polyclinic S. Orsola-Malpighi, Department of Organ Impairment and Transplants, Operative Unit of Infectious Diseases, Bologna
  - University Polyclinic Hospital of Modena, Department of General and Specialist Surgery, Operative Unit of Anesthesia and Intensive Care I, Modena
  - University Hospital of Pisa, Department of Gastroenterology and Infectious Diseases, Operative Unit of Infectious Diseases, Pisa
  - University Polyclinic Agostino Gemelli, Complex Operative Unit of Infectious Diseases 2, Rome
  - Hospital Maggiore University Hospital Ospedali Riuniti of Trieste Dept of ID, Trieste
  - University Hospital "Santa Maria della Misericordia" of Udine, Department of Specialist Medicine, Clinic of Infectious Diseases, Udine
- Romania (4):
  - Craiova County Emergency Clinical Hospital, ATI Clinic, Craiova, Dolj
  - Institute of Infectious Diseases, Bucharest, Sector 2
  - Pius Brinzeu County Emergency Clinical Hospital, Anesthesia and Intensive Care Department (Romania), Timișoara, Timiș County
  - Sfanta Parascheva Parascheva Iasi Clinical Hospital for Infectious Diseases, Iași
- Russia (3):
  - Kuban State Medical University, Krasnodar
  - Territorial Clinical Hospital, Krasnoyarsk
  - Mariinskaya City Hospital, Saint Petersburg
- Spain (12):
  - University Hospital Vall d'Hebron (HUVH), Department of Infectious Diseases, Barcelona, Catalonia
  - Hospital Clinic i Provincial de Barcelona, Department of Infectious Diseases, Barcelona, Catalonia
  - University Hospital Cruces, Unit of Infectious Diseases, Barakaldo
  - Hospital del Mar, Department of Infectious Diseases, Barcelona
  - General University Hospital Gregorio Maranon, Madrid
  - University Hospital Ramon y Cajal, Madrid
  - University Hospital Clinical San Carlos, Madrid
  - University Hospital La Paz, Madrid
  - University Hospital Virgen Macarena, Seville
  - University Hospital Nuestra Senora de Valme,, Seville
  - University Hospital Virgen del Rocio (HUVR), Seville
  - University Hospital La Fe, Valencia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Honore PM, Bassetti M, Cornely OA, Dupont H, Fortun J, Kollef MH, Pappas P, Pullman J, Vazquez J, Bielicka I, Dickerson S, Manamley N, Sandison T, Thompson GR. Length of hospital and intensive care unit stay in patients with invasive candidiasis and/or candidemia treated with rezafungin: a pooled analysis of two randomised controlled trials. Crit Care. 2024 Nov 11;28(1):361. doi: 10.1186/s13054-024-05152-2. PMID 39529079
- [Derived] Honore PM, Girardis M, Kollef M, Cornely OA, Thompson GR 3rd, Bassetti M, Soriano A, Huang H, Vazquez J, Kullberg BJ, Pappas PG, Manamley N, Sandison T, Pullman J, Nseir S. Rezafungin versus caspofungin for patients with candidaemia or invasive candidiasis in the intensive care unit: pooled analyses of the ReSTORE and STRIVE randomised trials. Crit Care. 2024 Oct 28;28(1):348. doi: 10.1186/s13054-024-05117-5. PMID 39468640
- [Derived] Smith HL, Bensman TJ, Mishra S, Li X, Dixon CA, Sheikh J, McMaster OG, Joshi A, Rubin DB, Goodwin A, Miller TJ, Danielsen ZY, Syed I, Shukla SJ, Iarikov D, Kim PW, Farley JJ. Regulatory Considerations in the Approval of Rezafungin (Rezzayo) for the Treatment of Candidemia and Invasive Candidiasis in Adults. J Infect Dis. 2024 Aug 16;230(2):505-513. doi: 10.1093/infdis/jiae146. PMID 38502709
- [Derived] Thompson GR 3rd, Soriano A, Honore PM, Bassetti M, Cornely OA, Kollef M, Kullberg BJ, Pullman J, Hites M, Fortun J, Horcajada JP, Kotanidou A, Das AF, Sandison T, Aram JA, Vazquez JA, Pappas PG. Efficacy and safety of rezafungin and caspofungin in candidaemia and invasive candidiasis: pooled data from two prospective randomised controlled trials. Lancet Infect Dis. 2024 Mar;24(3):319-328. doi: 10.1016/S1473-3099(23)00551-0. Epub 2023 Nov 23. PMID 38008099
- [Derived] Thompson GR, Soriano A, Skoutelis A, Vazquez JA, Honore PM, Horcajada JP, Spapen H, Bassetti M, Ostrosky-Zeichner L, Das AF, Viani RM, Sandison T, Pappas PG. Rezafungin Versus Caspofungin in a Phase 2, Randomized, Double-blind Study for the Treatment of Candidemia and Invasive Candidiasis: The STRIVE Trial. Clin Infect Dis. 2021 Dec 6;73(11):e3647-e3655. doi: 10.1093/cid/ciaa1380. PMID 32955088

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: Subjects in the CD101 IV treatment group 1 (Part A Only - up to 30 mITT subjects) will receive CD101 IV 400 mg on Day 1 and Day 8, with an optional dose of 400 mg on Day 15 (for all subjects) and an optional dose of 400 mg on Day 22 (only for subjects with IC), if needed.
  Daily intravenous placebo infusion when not administered CD101. Daily oral placebo as step down.
  CD101: Intravenous antifungal therapy
  intravenous placebo: normal saline
  oral placebo: microcrystalline cellulose
- Group 2: Subjects in the CD101 IV treatment group 2 (Part B Only - up to 30 mITT subjects) will receive CD101 IV 400 mg on Day 1 and Day 8, with an optional dose of 200 mg on Day 15 (for all subjects) and an optional dose of 200 mg on Day 22 (only for subjects with IC), if needed.
  Daily intravenous placebo infusion when not administered CD101. Daily oral placebo as step down.
  CD101: Intravenous antifungal therapy
  intravenous placebo: normal saline
  oral placebo: microcrystalline cellulose
- Group 3: Subjects in the caspofungin group will receive IV caspofungin (a single 70 mg loading dose on Day 1 followed by 50 mg once daily) for ≥3 days up to a maximum of 21 days for subjects with candidemia only and up to a maximum of 28 days for subjects with IC (with or without candidemia).
  After ≥3 days of IV therapy, subjects in the caspofungin group can be switched to oral step-down therapy of fluconazole (a loading dose of 800 mg [4 capsules] on the first day followed by 400 mg [2 capsules]/day thereafter). After switch to oral step down before Day 8, subjects in the caspofungin group will receive IV placebo on Day 8 to preserve the study blind.
  Caspofungin: Intravenous antifungal therapy
  Fluconazole: oral antifungal therapy
  intravenous placebo: normal saline
Period: Part A
Arm/Group | Group 1 | Group 2 | Group 3
Started (The Intent-to-Treat (ITT) population analyzed consisted of all subjects randomized to treatment. Subjects were analyzed based on the treatment group to which they were randomized. In Part A, subjects were randomized in a 1:1:1 ratio to receive rezafungin treatment Group 1, rezafungin Treatment Group 2 (defined below), or IV caspofungin Group 3. Enrollment into Part A closed and Part B began.) | 35 | 36 | 36
Completed | 23 | 28 | 22
Not Completed | 12 | 8 | 14
Not completed — Death | 3 | 4 | 6
Not completed — Lost to Follow-up | 2 | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1 | 2
Not completed — Physician Decision | 2 | 0 | 1
Not completed — Adverse Event | 2 | 0 | 1
Not completed — Noncompliance | 1 | 1 | 0
Not completed — Other | 1 | 1 | 3
Period: Part B
Arm/Group | Group 1 | Group 2 | Group 3
Started (The Intent-to-Treat (ITT) population analyzed consisted of all subjects randomized to treatment. Subjects were analyzed based on the treatment group to which they were randomized. In Part B, subjects were randomized 2:1 to receive rezafungin treatment or IV caspofungin.) | 46 | 21 | 33
Completed | 33 | 14 | 28
Not Completed | 13 | 7 | 5
Not completed — Death | 8 | 3 | 5
Not completed — Lost to Follow-up | 2 | 2 | 0
Not completed — Withdrawal by Subject | 3 | 1 | 0
Not completed — Other | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Intent-to-Treat (ITT) population analyzed consisted of all subjects randomized to treatment. Subjects were analyzed based on the treatment group to which they were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Group 3 | Total
Number analyzed (Participants) | 81 | 57 | 69 | 207
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 49 | 32 | 40 | 121
  >=65 years | 32 | 25 | 29 | 86
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.4 (15.86) | 60.0 (15.90) | 59.4 (15.85) | 59.6 (15.79)
Age, Continuous [Median (Full Range); unit: years] | 61.0 [24.0 to 88.0] | 63.0 [24.0 to 91.0] | 63.0 [24.0 to 93.0] | 62.0 [24.0 to 93.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 21 | 31 | 89
  Male | 44 | 36 | 38 | 118
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 9 | 7 | 24
  Not Hispanic or Latino | 73 | 46 | 59 | 178
  Unknown or Not Reported | 0 | 2 | 3 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 8 | 7 | 4 | 19
  White | 69 | 44 | 59 | 172
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 4 | 5 | 3 | 12
Region of Enrollment [Number; unit: participants]
  Greece | 6 | 6 | 8 | 20
  Canada | 1 | 1 | 3 | 5
  Romania | 2 | 0 | 3 | 5
  Belgium | 9 | 9 | 12 | 30
  Hungary | 2 | 0 | 0 | 2
  United States | 26 | 22 | 23 | 71
  Italy | 7 | 2 | 5 | 14
  Bulgaria | 4 | 1 | 2 | 7
  Russia | 2 | 1 | 0 | 3
  Spain | 22 | 15 | 13 | 50
Diagnosis [Count of Participants; unit: Participants]
  Candidemia | 62 | 46 | 56 | 164
  Invasive Candidiasis | 19 | 11 | 13 | 43
Estimated Normalized Creatinine Clearance [Mean (Standard Deviation); unit: mL/min/1.73m^2] — Population: Data was not captured at baseline for all subjects, preventing calculation of the normalized creatinine clearance.
  mL/min/1.73m^2
    number analyzed (Participants) | 79 | 50 | 64 | 193
    (all) | 90.8 (52.03) | 72.8 (52.14) | 87.1 (59.29) | 84.9 (54.78)
Estimated Normalized Creatinine Clearance [Median (Full Range); unit: mL/min/1.73m^2] — Population: Data was not captured at baseline for all subjects, preventing calculation of the normalized creatinine clearance.
  mL/min/1.73m^2
    number analyzed (Participants) | 79 | 50 | 64 | 193
    (all) | 81.8 [8.1 to 255.4] | 57.7 [5.9 to 294.7] | 74.4 [7.7 to 278.8] | 74.8 [5.9 to 294.7]
Acute Physiology and Chronic Health Evaluation (APACHE) II Score [Mean (Standard Deviation); unit: units on a scale] — The APACHE II score is a validated predictor of mortality in critically ill patients. It can be used as a surrogate measure for severity of illness in a patient and can be used in clinical trials at baseline to estimate the overall severity of illness in a patient population.
  Knaus WA, Draper EA, Wagner DP, Zimmerman JE. APACHE II: a severity of disease classification system. Critical Care Medicine 1985 13(10):818-29.
  APACHE II score = acute physiology score + age points + chronic health points. Minimum score = 0; maximum score = 71. Population: Data was not captured for all subjects, as some subjects did not have the APACHE II calculation performed.
  units on a scale
    number analyzed (Participants) | 79 | 55 | 63 | 197
    (all) | 13.4 (7.13) | 14.1 (6.72) | 14.0 (7.39) | 13.8 (7.07)
Acute Physiology and Chronic Health Evaluation (APACHE) II Score [Median (Full Range); unit: units on a scale] — The APACHE II score is a validated predictor of mortality in critically ill patients. It can be used as a surrogate measure for severity of illness in a patient and can be used in clinical trials at baseline to estimate the overall severity of illness in a patient population.
  Knaus WA, Draper EA, Wagner DP, Zimmerman JE. APACHE II: a severity of disease classification system. Critical Care Medicine 1985 13(10):818-29.
  APACHE II score = acute physiology score + age points + chronic health points. Minimum score = 0; maximum score = 71. Population: Data was not captured for all subjects, as some subjects did not have the APACHE II calculation performed.
  units on a scale
    number analyzed (Participants) | 79 | 55 | 63 | 197
    (all) | 12.0 [2.0 to 31.0] | 14.0 [2.0 to 28.0] | 13.0 [1.0 to 35.0] | 12.0 [1.0 to 35.0]
Acute Physiology and Chronic Health Evaluation (APACHE) II Category [Count of Participants; unit: Participants] — The APACHE II score is a validated predictor of mortality in critically ill patients. It can be used as a surrogate measure for severity of illness in a patient and can be used in clinical trials at baseline to estimate the overall severity of illness in a patient population.
  Knaus WA, Draper EA, Wagner DP, Zimmerman JE. APACHE II: a severity of disease classification system. Critical Care Medicine 1985 13(10):818-29.
  APACHE II score = acute physiology score + age points + chronic health points. Minimum score = 0; maximum score = 71.
  Participants
    0-9 | 23 | 15 | 17 | 55
    10-19 | 39 | 26 | 37 | 102
    ≥20 | 17 | 14 | 9 | 40
    Missing | 2 | 2 | 6 | 10

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Treatment Emergent Adverse Events [Safety and Tolerability]
Description: Number of Subjects with Incidence of Treatment Emergent Adverse Events based on clinical chemistry, hematology and urine analysis laboratory test, vital sign, physical exams and ECG abnormalities.
Time Frame: From first dose of study drug through Days 45-52 for subjects with candidemia only or Days 52-59 for subjects with IC, with or without candidemia.
Population: Safety Population includes all subjects randomized to treatment and who received any amount of study drug. A total of 202 subjects were included in the Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 81 | 53 | 68
Participants | 71 | 49 | 55

2. Primary Outcome: Resolution of Systemic Signs Attributable to Candidemia and/or Invasive Candidiasis and Mycological Eradication [Overall Success]
Description: Number of subjects with mycological eradication and complete resolution of all systemic signs of candidemia and/or invasive candidiasis which were present at baseline
Time Frame: Day 14 (± 1 day)
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 76 | 46 | 61
Participants | 46 | 35 | 41

3. Secondary Outcome: Mycological Eradication and Resolution of Systemic Signs
Description: Evaluate overall success signs (mycological eradication and resolution of systemic signs attributable to candidemia and/or IC) in the mITT population.
Time Frame: Day 5, and Follow-up (FU Days 45-52 for subjects with candidemia only or Days 52-59 for subjects with IC, with or without candidemia.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 76 | 46 | 61
Participants
  Day 5 | 42 | 34 | 34
  Follow-up | 36 | 30 | 36

4. Secondary Outcome: Mycological Eradication
Description: Evaluate mycological success (eradication) in the mITT population.
Time Frame: Day 5, Day 14 (±1 day), and FU (Days 45-52 for subjects with candidemia only or Days 52-59 for subjects with IC, with or without candidemia)
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 76 | 46 | 61
Participants
  Day 5 | 50 | 35 | 38
  Day 14 | 50 | 35 | 42
  Follow-up | 39 | 30 | 36

5. Secondary Outcome: Clinical Cure
Description: Evaluate clinical cure as assessed by the Investigator in the mITT population. Subjects must meet all of the following requirements:
  * Resolution of attributable systemic signs and symptoms of candidemia/IC that were present at baseline
  * No new systemic signs or symptoms attributable to candidemia/IC
  * No additional systemic antifungal therapy administered for candidemia/IC
  * The subject is alive
Time Frame: Day 14 (±1 day) and FU (Days 45-52 for subjects with candidemia only or Days 52-59 for subjects with IC, with or without candidemia).
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 76 | 46 | 61
Participants
  Day 14 | 53 | 37 | 43
  Follow-up | 42 | 32 | 38

6. Secondary Outcome: Evaluate PK (Cmax)
Description: Evaluate maximum plasma concentration (Cmax) (Part A only)
Time Frame: Day 1, 10 minutes before end of infusion (EOI)
Population: PK Population: all rezafungin-treated subjects from Part A with at least 1 plasma sample obtained for PK analysis.
Measure: Mean (Standard Deviation); unit: μg/mL
Groups:
- Group 2: Subjects in the CD101 IV treatment group 1 (Part A Only - up to 30 mITT subjects) will receive CD101 IV 400 mg on Day 1 and Day 8, with an optional dose of 400 mg on Day 15 (for all subjects) and an optional dose of 400 mg on Day 22 (only for subjects with IC), if needed.
  Daily intravenous placebo infusion when not administered CD101. Daily oral placebo as step down.
  CD101: Intravenous antifungal therapy
  intravenous placebo: normal saline
  oral placebo: microcrystalline cellulose
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 29 | 30
μg/mL | 15.258 (5.5430) | 14.743 (5.6450)

7. Secondary Outcome: Evaluate PK (Cmin)
Description: Evaluate minimum plasma concentration (Cmin) (Part A only)
Time Frame: Day 8, predose
Population: PK Population: all rezafungin-treated subjects from Part A with at least 1 plasma sample obtained for PK analysis.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 25 | 28
μg/mL | 2.050 (0.9767) | 2.313 (1.2165)

8. Secondary Outcome: Evaluate PK (Cmin)
Description: Evaluate minimum plasma concentration (Cmin) (Part A only)
Time Frame: Day 15, predose
Population: PK Population: all rezafungin-treated subjects from Part A with at least 1 plasma sample obtained for PK analysis.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 21 | 21
μg/mL | 3.068 (1.4565) | 2.131 (0.8506)

ADVERSE EVENTS:
Time Frame: Adverse events were collected following the signing of the informed consent at screening and throughout the study until the follow up visit (Days 45-52 for subjects with candidemia only or Days 52-59 for subjects with IC, with or without candidemia).
Description: All-Cause Mortality was assessed in the Intent-to-Treat (ITT) Population. The ITT Population consisted of all subjects randomized to treatment. Serious and Other Adverse Events were assessed in the Safety Population. The Safety Population consisted of all subjects randomized who received any amount of study drug. All safety analyses were performed by actual treatment received.
Arm/Group | Group 1 | Group 2 | Group 3
All-Cause Mortality (participants affected / at risk) | 14/81 | 7/57 | 13/69
Serious Adverse Events (participants affected / at risk) | 35/81 | 28/53 | 29/68
Other Adverse Events (participants affected / at risk) | 70/81 | 49/53 | 53/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (N=81) | Group 2 (N=53) | Group 3 (N=68)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0 | 0
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Sickle cell anaemia with crisis (Blood and lymphatic system disorders) | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 1 | 0 | 0
Atrial flutter (Cardiac disorders) | 1 | 0 | 0
Atrioventricular block (Cardiac disorders) | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1 | 1
Cardiac failure (Cardiac disorders) | 0 | 1 | 1
Right ventricular failure (Cardiac disorders) | 0 | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1
Colonic fistula (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 1 | 0
Haemorrhagic ascites (Gastrointestinal disorders) | 0 | 0 | 1
Impaired gastric emptying (Gastrointestinal disorders) | 1 | 0 | 0
Peritoneocutaneous fistula (Gastrointestinal disorders) | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
Generalised oedema (General disorders) | 0 | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 2 | 0 | 2
Biloma (Hepatobiliary disorders) | 0 | 1 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 0 | 0
Abdominal abscess (Infections and infestations) | 1 | 1 | 0
Abscess limb (Infections and infestations) | 1 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 2 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 1
Candida sepsis (Infections and infestations) | 0 | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 2 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 1
Endocarditis candida (Infections and infestations) | 0 | 0 | 1
Escherichia bacteraemia (Infections and infestations) | 0 | 1 | 0
Pelvic abscess (Infections and infestations) | 1 | 0 | 0
Peritonitis (Infections and infestations) | 1 | 0 | 0
Peritonitis bacterial (Infections and infestations) | 2 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 0 | 1
Pulmonary sepsis (Infections and infestations) | 0 | 0 | 1
Renal abscess (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 1 | 2 | 2
Septic embolus (Infections and infestations) | 0 | 1 | 0
Septic shock (Infections and infestations) | 9 | 1 | 2
Staphylococcal bacteraemia (Infections and infestations) | 0 | 2 | 0
Systemic candida (Infections and infestations) | 1 | 0 | 0
Urosepsis (Infections and infestations) | 1 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 0 | 0 | 1
Post procedural fistula (Injury, poisoning and procedural complications) | 1 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0
Tracheal haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 | 0 | 0
Aspiration bronchial (Investigations) | 0 | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Post transplant lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 1 | 0 | 0
Encephalopathy (Nervous system disorders) | 1 | 0 | 0
Metabolic encephalopathy (Nervous system disorders) | 1 | 0 | 0
Neurodegenerative disorder (Nervous system disorders) | 0 | 1 | 0
Neurological symptom (Nervous system disorders) | 0 | 1 | 0
Peroneal nerve palsy (Nervous system disorders) | 0 | 1 | 0
Seizure (Nervous system disorders) | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1
Henoch-Schonlein purpura (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Arterial haemorrhage (Vascular disorders) | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1
Shock (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (N=81) | Group 2 (N=53) | Group 3 (N=68)
Hypokalaemia (Metabolism and nutrition disorders) | 13 | 9 | 9
Diarrhoea (Gastrointestinal disorders) | 7 | 11 | 10
Vomiting (Gastrointestinal disorders) | 6 | 8 | 5
Pyrexia (General disorders) | 9 | 4 | 6
Anaemia (Blood and lymphatic system disorders) | 6 | 7 | 4
Nausea (Gastrointestinal disorders) | 4 | 8 | 6
Abdominal pain (Gastrointestinal disorders) | 5 | 5 | 4
Hypotension (Vascular disorders) | 6 | 2 | 4
Insomnia (Psychiatric disorders) | 4 | 4 | 2
Oedema peripheral (General disorders) | 6 | 2 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 4 | 3 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2018-04-20): https://cdn.clinicaltrials.gov/large-docs/62/NCT02734862/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-17): https://cdn.clinicaltrials.gov/large-docs/62/NCT02734862/SAP_001.pdf